CLINICAL TRIAL: NCT02598466
Title: Patient-Reported Efficacy of Subcutaneous Abatacept in Rheumatoid Arthritis: An Evaluation Of Patients In a Compassionate Use Programme in South Africa
Brief Title: Patient-Reported Efficacy of Subcutaneous (SC) Abatacept in Rheumatoid Arthritis (RA) - South Africa
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Hexor, South Africa (Other)
Responsible Party: Sponsor
Other Study IDs: IM101-572
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Abatacept
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept

SUMMARY:
Research question: what are the patterns of patient-reported changes in physical function among adult patients using SC abatacept with moderate to severe RA since commencement of the compassionate use program (CUP).

ELIGIBILITY:
Inclusion Criteria:

* The global clinical trials and associated long-term extension phases imposed inclusion and exclusion criteria. Only patients that completed the clinical trials and the long-term extension phase were eligible for inclusion in the CUP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Patterns of change in patient assessments of physical function with scores of the Health Assessment Questionnaire (HAQ) among users of SC Abatacept for RA since the commencement of a CUP in South Africa's private sector | Approximately 2 years

SECONDARY OUTCOMES:
Demographic characteristics (age, gender, education and population group) of patients | Approximately 2 years
Clinical characteristics (comorbidities including Tuberculosis, medication use, and adverse events) of patients | Approximately 2 years
Reasons for discontinuation based on the reasons mentioned in Questionnaire | Approximately 2 years
  Reasons for discontinuation: defined as common responses given for stopping treatment and include death, adverse event, lack of efficacy, lost to follow-up, withdrawal of consent, or other reasons
Reasons for skipping treatment based on the reasons mentioned in Questionnaire | Approximately 2 years
  Reasons for skipping treatment: defined as explanations given for inability to adhere to the recommended treatment regime and include fear of side effects, lack of access (too far) to medicine, inconvenient to use, too busy or forgetting, or other reasons
Association of demographic and clinical characteristics based on Standard Disability Index of the Health Assessment Questionnaire (HAQ-DI) scores | Approximately 2 years
Changes in physical functioning against clinical trial and long-term extension phase data based incidence of adverse events | Approximately 2 years
  Adverse events: defined as any untoward medical event in a patient whether related or unrelated to SC abatacept and may include any sign (laboratory finding), symptom, or disease

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx